CLINICAL TRIAL: NCT00370877
Title: Recombinant Human Activated Factor VII as Salvage Therapy in Women With Severe Postpartum Hemorrhage
Brief Title: rhuFVIIa in Post-partum Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: University Hospital, Lille (Other); Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Montpellier (Other); University Hospital, Geneva (Other); Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC-I/2005/GL-01; 2005-005801-40 (EudraCT Number)
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Postpartum Hemorrhage
Keywords: Post-partum hemorrhage; Arterial embolization; Surgery; Hysterectomy; Activated recombinant human factor VII
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — recombinant FVIIa; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care for post-partum hemorrhage (Active Comparator): The patients included in this arm of the study will recieve standard care for post-partum hemorrhage.
  Interventions: Procedure: Standard Care
- rFVIIa (Experimental): The patients included in this arm of the study will recieve standard care for post-partum hemorrhage plus a slow intravenous injection (2ml/min) of rFVIIa (60µg/kg)
  Interventions: Drug: rFVIIa

INTERVENTIONS:
Drug: rFVIIa — The patients included in this arm of the study will recieve standard care for post-partum hemorrhage plus a slow intravenous injection (2ml/min) of rFVIIa (60µg/kg)
  Other Names: Experimental; Novo 7; eptacog alpha (activated)
  Arms: rFVIIa
Procedure: Standard Care — Patients will recieve standard care for post partum hemorrhage according to current recommendations.
  Other Names: Standard
  Arms: Standard care for post-partum hemorrhage

SUMMARY:
The aim of this clinical research project is to evaluate the use of the recombinant human activated factor VII (rhFVIIa), given as a salvage therapy, in women with a dramatic postpartum hemorrhage still ongoing after all the currently available medical and surgical treatments. We are going to compare its early use, before elective surgery or arterial embolization, to its late use, after embolization or surgery, before salvage hysterectomy.

DETAILED DESCRIPTION:
Depending on the country and the publications, postpartum hemorrhage is either the first or the second cause of maternal death in the world, including developed countries. According to the WHO, it is responsible for twenty two percent of maternal deaths. In France, postpartum hemorrhage accounts for five percent of delivery complications. Three percent of them are severe, leading to uncontrolled bleeding which intensity is higher than 1000 ml of blood during the 24 hours following delivery. In France, they are involved in 20 new deaths per year; it is the first cause of maternal mortality. Indeed, it remains a significant source of morbidity: severe anaemia, blood transfusion, transfusion complications, acquired coagulation disorders and hemostatic hysterectomy.

There are two different types of postpartum hemorrhage: early and late hemorrhages. Early hemorrhages are more common and occur in the first 24H after delivery. Uterine atony is the main cause of early hemorrhage. However, visual assessment underestimates the amount of blood loss in around forty five percent of cases. Emergency treatment is therefore sometimes undertaken with some delay, giving time for disseminated intravascular coagulation (DIC) to occur, which worsens the prognosis. They are usually treated by medical resuscitation, blood transfusion, selective arterial embolisation and finally hysterectomy in case of ongoing uncontrolled bleeding. Medical treatment and obstetric manoeuvres are usually effective. Artificial delivery of the placenta should be performed immediately if the placenta is incomplete. Afterwards, oxytocin and prostaglandin derivatives are given. At the same time, anemia and hemostatic abnormalities are treated by transfusion of fresh frozen plasma and packed cells. When the measures are insufficient, surgery is necessary. Bilateral ligation of hypogastric arteries or controlled embolisation is recommended. In the case of uncontrolled bleeding, hemostatic hysterectomy is performed as a salvage therapy. Also, the efficacy of ligation of the hypogastric arteries remains controversial. Therefore, the success rate of ligation of the hypogastric arteries is only forty two percent, so that in many cases hysterectomy is required, which induces a definitive sterility. The development of interventional radiology has offered a new approach for the management of postpartum hemorrhage. Many publications have showed the usefulness of the procedure, whose success rate is around ninety percent. However, a specific technical plateau is needed, which is far to be available at any place and at any moment. For patients delivering far away from these technical sites, limiting blood loss is crucial. Among the methods aiming at limiting obstetrical hemorrhage, special concern was given to recombinant activated factor VII, a drug used with good therapeutic results in symptomatic patients with hemophilia and inhibitors. It has already been applied in interventions situations.

Taking into consideration the above described aspects, our goal is thus to evaluate the potential medical interest of giving rhFVIIa early in the course of hemorrhage, compared to giving it as a salvage therapy after arterial selective embolization or hysterectomy in patients still bleeding, in order to avoid hemostatic hysterectomy.

In the literature, IV infusion of rFVIIa stopped ongoing diffuse hemorrhage, rapidly, and no further transfusion was required after rFVIIa injection. Then rFVIIa, might be a strong complementary agent in the management of major postpartum hemorrhage. Optimal dose, timing and safety characteristics of rFVIIa administration remain to be determined.

Therefore, the main objectives of the study are:

1. to evaluate the reduction of the absolute risk of arterial embolization/surgery/hysterectomy in patients receiving a unique early infusion of rhuFVIIa (60 µg/kg body weight);
2. to evaluate the number of women necessary to treat to avoid one arterial embolization/surgery/hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Severe postpartum hemorrhage, i.e non responsive to sulprostone infusion

Exclusion Criteria:

* < 18 years
* personal antecedent of arterial or venous thrombosis
* written informed consent not approved/signed by the patient or her husband

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2007-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Clinical parameters: intensity of the hemorrhage, before and one hour after the end of the rhuFVIIa infusion (use of a graduated blood collector bag device). | 1 hour
Any transfusion (number of units and volume) of red blood cells, platelet or fresh frozen plasma. Haemodynamics-related parameters (non-invasive arterial pressure,heart rate, diuresis,..). | 7 Hours
Biological parameters:packed red cell volume, hemoglobin, etc. | 12 hours
Therapeutic interventions aiming at controlling postpartum hemorrhage: selective arterial embolization, ligation of hypogastric arteries, hysterectomy. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Gris, MD, PhD, Study Director — University Hospital, Nimes, France
Locations (8):
- France (7):
  - University Hospital, Lille, Lille, Lille
  - University Hospital of Montpellier, Montpellier, Montpellier
  - University Hospital, Nice, Nice, Nice
  - Hôpital Antoine Béclère -APHP, Clamart
  - Laboratoire d'hématologie, Groupe Hospitalo-Universitaire Caremeau, Nîmes
  - Centre Hospital University of Nimes, Nîmes
  - Maternite CHU de Cochin - APHP, Paris
- University Hospital, Geneva, Geneva, Switzerland

REFERENCES:
- [Derived] Lavigne-Lissalde G, Aya AG, Mercier FJ, Roger-Christoph S, Chauleur C, Morau E, Ducloy-Bouthors AS, Mignon A, Raucoules M, Bongain A, Boehlen F, de Moerloose P, Bouvet S, Fabbro-Peray P, Gris JC. Recombinant human FVIIa for reducing the need for invasive second-line therapies in severe refractory postpartum hemorrhage: a multicenter, randomized, open controlled trial. J Thromb Haemost. 2015 Apr;13(4):520-9. doi: 10.1111/jth.12844. Epub 2015 Mar 11. PMID 25594352